CLINICAL TRIAL: NCT00803634
Title: A Safety and Efficacy Study of Blood Pressure Control in Acute Heart Failure - A Pilot Study (PRONTO)
Brief Title: Clevidipine in the Treatment of Blood Pressure in Patients With Acute Heart Failure (PRONTO)
Acronym: PRONTO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC-CLV-08-01; TMC-CLV-08-01 (Other: Sponsor)
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension; Heart Failure
Keywords: Hypertension; Antihypertensive Agent; Calcium Channel Blocker
MeSH Terms: conditions — Hypertension; Heart Failure | interventions — clevidipine; Nitroglycerin; Nicardipine; Nitroprusside; Isosorbide Dinitrate; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clevidipine (Experimental): Clevidipine (0.5 mg/mL in 20% lipid emulsion) was administered intravenously via a single dedicated line to all patients randomized to the clevidipine arm. Clevidipine was infused at an initial rate of 2 mg/h for the first 3 minutes. If blood pressure was not in the target range at 3 minutes, clevidipine was titrated to effect thereafter by doubling the dose every 3 min, per physician discretion and as tolerated by the patient until the desired effect until the SBP target range was attained. Once target range was achieved, the infusion rate could be increased or decreased as needed to maintain blood pressure for minimum of 30 minutes and a maximum duration of 96 hours. The minimum infusion rate was 1 mg/h and maximum infusion rate was 32 mg/h.
  Interventions: Drug: Clevidipine
- Standard of Care IV antihypertensive (Active Comparator): For patients randomized to standard of care (SOC) IV antihypertensive treatment, a continuous infusion of an intravenous antihypertensive agent represented standard of care. The selection of treatment was at the discretion of the investigator. The infusion was to be administered according to the institution's treatment practice.
  Interventions: Drug: Standard of Care IV antihypertensive

INTERVENTIONS:
Drug: Clevidipine — Clevidipine was to be administered continuously as monotherapy during the first 30 minutes. Use of an alternative IV antihypertensive agent(s) was discouraged and was limited to where medically necessary to maintain patient safety. Patients who received an alternative antihypertensive agent along with the study drug were allowed to continue in the study. If transition to an oral antihypertensive agent was required, it was to be administered approximately 1 hour prior to the termination of clevidipine with study drug down-titrated or terminated in order to maintain the desired blood pressure level.
  Other Names: Cleviprex; clevidipine emulsion; clevidipine injectible emulsion
  Arms: Clevidipine
Drug: Standard of Care IV antihypertensive — SOC IV antihypertensive agent will be administered for a minimum of 30 min and, if medically warranted, may continue beyond 96 hours at the investigator's discretion. As with clevidipine, the SOC agent was to be administered continuously as monotherapy during the first 30 minutes. Use of an alternative agent(s) was discouraged and was limited to where medically necessary to maintain patient safety. Higher dose titration rates were required to be attempted prior to making the decision to switch to or add on an alternative antihypertensive agent(s). Patients who received an alternative antihypertensive agent with SOC were allowed to continue in the study. If transition to an oral antihypertensive agent was required, it was to be administered per institutional practice.
  Other Names: nitroglycerin; nicardipine; sodium nitroprusside; isosorbide dinitrate; hydralizine; diltiazem
  Arms: Standard of Care IV antihypertensive

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of intravenous (IV) clevidipine as compared with standard of care IV antihypertensive agents for blood pressure (BP) lowering in patients with acute heart failure and elevated BP.

DETAILED DESCRIPTION:
This study was an open-label randomized efficacy and safety pilot trial in patients with acute heart failure (AHF) and hypertension (systolic blood pressure [SBP] ≥160 mm Hg) requiring parenteral antihypertensive therapy. Eligible patients were randomized to receive clevidipine or standard of care (SOC) intravenous antihypertensive treatment in an open-label manner in a ratio of 1:1. At the time of randomization, a patient-specific, prespecified SBP target range was determined and be recorded, prior to study drug treatment. Information on the dosing regimen, use of additional or alternative agents and transition to oral therapy if needed is detailed in the study 'ARM' and 'INTERVENTION' sections.

A Data Safety Monitoring Board was utilized periodically throughout the study to monitor the safety of patients. Adverse events were assessed for 7 days post-study randomization or hospital discharge, whichever occured first. Serious adverse events (SAEs) were assessed for 30 days following study randomization. Subjects were contacted by telephone or in person up to 5 days after their 30-day time point to determine if any SAEs occurred following study drug treatment and to follow up on the Heath Economic assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Presentation consistent with acute heart failure and pulmonary congestion on physical examination as evidenced by rales
* Baseline systolic blood pressure (immediately prior to initiation of study drug) of ≥160 mm Hg
* Dyspnea score (sitting) of at least 5 on a 10 cm visual analog scale (VAS)
* Required IV antihypertensive therapy to lower blood pressure
* Written informed consent

Exclusion Criteria:

* Administration of an agent (IV or oral) for the treatment of elevated BP within the previous 2 hours of randomization. (Previous short-acting non-IV nitrates, continuous positive airway pressure (CPAP), and bi-level positive airway pressure (BiPAP) were permitted)
* Chest pain and/or electrocardiogram with ST segment changes consistent with acute coronary syndrome
* Known or suspected aortic dissection
* Acute myocardial infarction within the prior 14 days
* Dialysis-dependant renal failure
* Requirement for immediate endotracheal intubation
* Positive pregnancy test, known pregnancy or breast feeding female
* Intolerance or allergy to calcium channel blockers
* Allergy to soybean oil or egg lecithin
* Known liver failure, cirrhosis or pancreatitis
* Prior directives against advanced life support
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2008-12; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Frank Peacock, MD, Principal Investigator — The Cleveland Clinic
Locations (13):
- United States (9):
  - Jackson Hospital, Montgomery, Alabama
  - Centinela Hospital, Inglewood, California
  - Louisiana State University Health Sciences Center, Baton Rouge, Louisiana
  - Louisiana State University Health Sciences Center - Emergency Medicine, New Orleans, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - Stony Brook University and Medical Center, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
- France (3):
  - Hopial AP-HP Hotel-Dieu, Paris
  - Hopital AP-HP La Pitie Sapetriere, Paris
  - Hopital AP-HP Lariboisiere Urgencies-SMUR, Paris
- Charité - Universitätsmedizin Berlin, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with symptoms of acute heart failure (AHF) and elevated blood pressure (BP) presented to the Emergency Departments at 13 hospitals (9 US; 3 France; 1 Germany) between Feb 2009 and Feb 2012 and received either clevidipine or standard of care (SOC) continuous IV antihypertensive therapy for management of their blood pressure.
Pre-assignment Details: Eligible patients who met all inclusion and none of the exclusion criteria, including confirmation that systolic blood pressure (SBP) was ≥160 mm Hg immediately prior to study drug, were randomized into the study. If SBP < 160 mm Hg immediately prior to drug, the patient was not to receive study drug and was treated per institutional practice.
Groups:
- Clevidipine: Clevidipine (0.5 mg/mL in 20% lipid emulsion) was administered intravenously via a single dedicated line to all patients randomized to the clevidipine arm. Clevidipine was titrated to effect thereafter by doubling the dose every 3 minutes, per physician discretion and as tolerated by the patient, until the desired SBP target range was attained. The infusion rate could then be increased or decreased as needed in order to maintain blood pressure for minimum of 30 minutes and a maximum duration of 96 hours. The minimum infusion rate was 1 mg/h and maximum infusion rate was 32 mg/h.
- Standard of Care: The selection of the standard of care (SOC) IV antihypertensive treatment agent was at the discretion of the investigator. The infusion was administered per the institution's treatment practice. Dose titrations were to be performed to the maximum allowed or tolerated dose in order to achieve SBP control within the patient-specified SBP target range within the first 30 minutes. SOC was to be administered for a minimum of 30 minutes and, if medically warranted, could continue beyond 96 hours at the investigator's discretion.
Period: Overall Study
Arm/Group | Clevidipine | Standard of Care
Started | 51 (All patients dosed with clevidipine [Safety population]) | 53 (All patients dosed with SOC antihypertensive therapy [Safety population])
mITT (Dosed & Have Confirmed AHF) | 44 (All patients dosed with clevidipine and confirmed to have AHF [mITT population]) | 41 (All patients dosed with SOC antihypertensive therapy and confirmed to have AHF [mITT population])
Completed | 45 (All patients dosed with clevidipine [Safety population]) | 48 (All patients dosed with SOC antihypertensive therapy [Safety population])
Not Completed | 6 | 5
Not completed — Withdrew Consent | 1 | 0
Not completed — Lost to Follow-up | 2 | 3
Not completed — Death | 3 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population: Includes all patients dosed with clevidipine (for patients randomized to the clevidipine arm) of standard of care (SOC) (for patients randomized to the SOC arm) continuous IV antihypertensive therapy.
Groups:
- Clevidipine Emulsion: All randomized and eligible patients who received any dose of clevidipine.
- SOC IV Antihypertensive Therapy: All randomized and eligible patients who received any SOC dose.
- Total: Total of all reporting groups
Arm/Group | Clevidipine Emulsion | SOC IV Antihypertensive Therapy | Total
Number analyzed (Participants) | 51 | 53 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (14.95) | 60.2 (14.89) | 61.0 (14.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 54
  Male | 26 | 24 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 50 | 53 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 44 | 83
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mm Hg] | 188.2 (25.02) | 184.8 (21.92) | 186.5 (23.44)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mm Hg] | 102.2 (24.14) | 99.2 (24.28) | 100.7 (24.14)

OUTCOME MEASURES:

1. Primary Outcome: Time to First Achieve Initial Prespecified SBP Target Range and 15% Reduction From Baseline Within First 30 Minutes
Description: Time to first achieve the initial pre-specified systolic blood pressure (SBP) target range and a 15% SBP reduction from baseline is the time in minutes between the initiation of study medication and the time the patient first achieved both components. Median time was estimated using Kaplan Meier method. 95% two-sided confidence interval of the median time is from 'Simon and Lee, 1982'. If patients did not reach both components within 30 minutes from the initial treatment with study medication, or another antihypertensive agent was administered, the patient was censored at 30 minutes or the time when another antihypertensive agent is given, whichever came first.
Time Frame: Initiation of study drug through the initial 30-minutes
Population: mITT population: All randomized and eligible patients who were dosed with study drug and have a baseline SBP ≥160 mm Hg, at least one post-baseline on-treatment SBP measurement, and a confirmed diagnosis of AHF
Measure: Median (95% Confidence Interval); unit: Minutes
Groups:
- Clevidipine: Clevidipine was titrated to effect thereafter by doubling the dose every 3 minutes, per physician discretion and as tolerated by the patient, until the desired SBP target range was attained. The infusion rate could then be increased or decreased as needed in order to maintain blood pressure for minimum of 30 minutes and a maximum duration of 96 hours. The minimum infusion rate was 1 mg/h and maximum infusion rate was 32 mg/h.
Arm/Group | Clevidipine | Standard of Care
Number analyzed (Participants) | 44 | 41
Minutes | 15.0 [15.0 to 21.0] | NA [NA to NA] — NA=Not Reached: Median time to achieve this goal could not be determined in the SOC IV therapy group because less than 50% (15/41; 36.6%) of patients achieved both the pre-specified target range and a 15% reduction in SBP within the first 30 minutes.

2. Secondary Outcome: Percentage Reaching Prespecified Target Range Without Falling Below Lower Limit of Target Range Within First 30 Minutes
Description: The percentage of patients reaching this endpoint was calculated within each treatment group using the number of mITT patients reaching the endpoint divided by the number of mITT patients, and multiplied by 100. Two-tailed 95% CIs were computed for these percentages.
Time Frame: Initiation of study drug through the initial 30-minutes
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- SOC IV Therapy: The selection of the standard of care (SOC) IV antihypertensive treatment agent was at the discretion of the investigator. The infusion was administered per the institution's treatment practice. Dose titrations were to be performed to the maximum allowed or tolerated dose in order to achieve SBP control within the patient-specified SBP target range within the first 30 minutes. SOC was to be administered for a minimum of 30 minutes and, if medically warranted, could continue beyond 96 hours at the investigator's discretion.
Arm/Group | Clevidipine | SOC IV Therapy
Number analyzed (Participants) | 44 | 41
Percentage of patients | 45.5 [30.7 to 60.2] | 51.2 [35.9 to 66.5]

3. Secondary Outcome: SBP Area Under the Curve (AUC) Outside Prespecified Target Range
Description: The magnitude and duration of SBP excursions was calculated as the area under the curve (AUC) for each patient, using the trapezoidal rule, related to time (in minutes) that each patient's SBP was outside the target range. AUC was determined based on data collected from the initiation of study medication through the end of monotherapy treatment up to 96 hours, normalized per hour, and expressed as mmHg × minute/hour.
Time Frame: Initiation of study drug through end of monotherapy (up to 96 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg x min/h
Arm/Group | Clevidipine | Standard of Care
Number analyzed (Participants) | 44 | 41
mm Hg x min/h | 494.96 (428.554) | 966.15 (860.278)

4. Secondary Outcome: Percentage Falling Below Lower Limit of SBP Target Range Within First 30 Minutes
Description: The percentage of patients in whom the SBP fell below the lower limit of the prespecified target range at any time during the first 30 minutes was calculated within each treatment group using the number of mITT patients achieving the endpoint divided by the number of mITT patients and multiplied by 100. Two-tailed 95% CIs were computed for these percentages.
Time Frame: Initiation of study drug through the initial 30-minutes
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Clevidipine | Standard of Care
Number analyzed (Participants) | 44 | 41
Percentage of patients | 34.1 [20.5 to 49.9] | 2.4 [0.1 to 12.9]

5. Secondary Outcome: Percentage Falling Below Lower Limit of SBP Target Range at Any Time During Study
Description: The percentage of patients in whom the SBP fell below the lower limit of the prespecified target range at any time during the entire study drug treatment period (up to 96 hours) was calculated within each treatment group using the number of mITT patients achieving the endpoint divided by the number of mITT patients and multiplied by 100. Two-tailed 95% CIs were computed for these percentages.
Time Frame: Initiation through termination of study drug (up to 96 hours)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Clevidipine | Standard of Care
Number analyzed (Participants) | 44 | 41
Percentage of patients | 68.2 [52.4 to 81.4] | 70.7 [54.5 to 83.9]

6. Secondary Outcome: Change From Baseline in Dyspnea (Measured By VAS) at Each Time Point
Description: A validated visual analog scale (VAS) with a horizontal ruler showing increments from 0 to 100 mm with 0 = Best and 100 = Worst was used. The test was asked from the patient's perspective and had to be administered with patient sitting. Relative change in VAS from baseline is the value at each time point minus the baseline value. Relative change from baseline was summarized descriptively (with associated two-tailed 95% CIs of the mean values) at 15, 30 and 45 minutes and at 1, 2, 3 hours and 12 hours, and 1 hour post termination of study drug treatment.
Time Frame: Baseline (immediately prior to study drug administration) through 1 hour after study drug termination
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Clevidipine | Standard of Care
Number analyzed (Participants) | 44 | 41
millimeters (mm)
  Baseline Through Initial 15 Min- CLV n=44;SOC n=38 | -18.6 (17.49) | -16.1 (19.78)
  Baseline Through Initial 30 Min- CLV n=43;SOC n=39 | -28.8 (19.94) | -22.8 (21.03)
  Baseline Through Initial 45 Min- CLV n=43;SOC n=39 | -37.1 (20.87) | -27.9 (21.73)
  Baseline Through Initial 1 H- CLV n=41;SOC n=38 | -43.6 (21.74) | -34.6 (23.38)
  Baseline Through Initial 2 H- CLV n=29;SOC n=29 | -45.2 (22.66) | -35.3 (22.30)
  Baseline Through Initial 3 H- CLV n=14;SOC n=22 | -47.9 (16.57) | -40.5 (21.69)
  Baseline Through Initial 12 H- CLV n=0;SOC n=7 | NA (NA) — All patients in the clevidipine arm either completed the study or dropped out by the 12 hour time point. | -57.9 (15.18)
  Baseline Through 1 H Post Drug- CLV n=41;SOC n=33 | -50.1 (23.22) | -50.1 (26.09)

7. Secondary Outcome: Time to Use Other IV Antihypertensives During the Study Drug Administration
Description: The length of time to use other IV antihypertensive agents was defined as the duration in hours from the initiation of study drug through the time when any other concomitant IV antihypertensive agent was administered, thus, representing the time period without use of any other concomitant IV antihypertensive agent. Median time to use other IV antihypertensive agents was obtained using Kaplan-Meier method. If a patient did not receive any concomitant IV antihypertensive during the 96-hour treatment period, this patient was considered censored at 96 hours. If study drug was stopped less than 96 hours and the patient has no concomitant IV antihypertensive agent, the patient was considered censored when study drug was stopped.
Time Frame: Initiation of study drug through any other concomitant IV antihypertensive agent administered, up to 96 hours
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Clevidipine | Standard of Care
Number analyzed (Participants) | 44 | 41
Hours | NA [NA to NA] — NA=Not estimable: Less than 50% of patients received a concomitant IV antihypertensive during study drug administration. | 5.7 [1.7 to NA] — The upper limit of the 95% CI could not be calculated according to Samon and Lee, 1982.

8. Secondary Outcome: Percentage of Patients Who Received Any Alternative IV Antihypertensive Drug at Any Time During Study Drug Treatment
Description: The percentage of patients who received any alternative IV antihypertensive drug at any time during the study drug treatment period (up to 96 hours) was calculated using mITT patients within each treatment group.
Time Frame: Initiation through termination of study drug (up to 96 hours)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Clevidipine | Standard of Care
Number analyzed (Participants) | 44 | 41
Percentage of patients | 15.9 [5.1 to 26.7] | 51.2 [35.9 to 66.5]

9. Secondary Outcome: Percentage of Patients With at Least One Episode of SBP < 90 mm Hg During Study Drug Administration (up to 96 Hours)
Description: The percent of patients with at least one episode of SBP <90 mm Hg was calculated as the number of mITT patients who had at least one episode of SBP<90 mm Hg during study drug administration up to 96 hours divided by mITT patients, and multiplied by 100 for each treatment group.
Time Frame: Initiation through termination of study drug (up to 96 hours)
Population: Safety population: All randomized and eligible patients who were dosed with study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Clevidipine | Standard of Care
Number analyzed (Participants) | 51 | 53
Percentage of patients | 5.9 [1.2 to 16.2] | 1.9 [0.0 to 10.1]

10. Secondary Outcome: Number of Patients That Require Intubation During Study Drug Administration up to 96 Hours
Description: The number of patients requiring intubation was calculated based on the total number of mITT patients.
Time Frame: Initiation through termination of study drug (up to 96 hours)
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Clevidipine | Standard of Care
Number analyzed (Participants) | 44 | 41
Patients | 0 | 0

11. Primary Outcome: Percentage to First Achieve Initial Prespecified SBP Target Range [≥20 mm Hg and ≤40 mm Hg Apart] and 15% Reduction From Baseline Within First 30 Minutes
Description: Analysis of the percentage of patients achieving both components of this composite endpoint (attainment of the initial prespecified SBP target range and a 15% reduction in SBP from baseline) was calculated within each treatment group using the number of mITT patients achieving the SBP reduction goal divided by the number of mITT patients, and multiplied by 100.
Time Frame: Initiation of study drug through the initial 30-minutes
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Clevidipine | Standard of Care
Number analyzed (Participants) | 44 | 41
Percentage of patients | 70.5 [57.0 to 83.9] | 36.6 [21.8 to 51.3]

ADVERSE EVENTS:
Time Frame: ▪ Non-serious Adverse Events (AEs) assessed up to 7 days following randomization or discharge whichever occurred first, regardless of causal relationship to the study drug ▪ Serious AEs (SAEs) assessed up to 30 days post-randomization into the study.
Description: AEs/SAEs were recorded in the electronic case report form (eCRF) by study personnel as a means of submitting required data to study Sponsor. The investigator was to complete an SAE Report (SAER) for each SAE regardless of causality by study medications, which was faxed to the Sponsor's safety vendor within 24 hours of when the SAE was recognized.
Arm/Group | Clevidipine | Standard of Care
Serious Adverse Events (participants affected / at risk) | 12/51 | 10/53
Other Adverse Events (participants affected / at risk) | 20/51 | 19/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clevidipine (N=51) | Standard of Care (N=53)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (4) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clevidipine (N=51) | Standard of Care (N=53)
Nausea (Gastrointestinal disorders) | 6 | 6
Headache (Nervous system disorders) | 11 | 13
Insomnia (Psychiatric disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After initial multicenter results communications are published, or after 12 months from study closure (whichever occurs first), sponsor can review results communications prior to submission and can embargo submissions for a period of 45 days from the time submitted to the sponsor for review, agreeing to resolve differences of opinion or interpretation through scientific debate. Sponsor can request further delay for an additional 90 days to file any patent applications if deemed necessary.